CLINICAL TRIAL: NCT04002258
Title: Prolactin Change and Its Effectors in Chinese Patients With Schizophrenia After Antipsychotics Treatment
Brief Title: Prolactin Change in Chinese Patients With Schizophrenia After Antipsychotics Treatment
Status: Completed | Type: Observational
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Principal Investigator, LI, Huafang, Director and Clinical Professor, Shanghai Mental Health Center
Other Study IDs: CRC2018DSJ01-2
Record Dates: First submitted 2019-03-26; First posted 2019-06-28 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Schizophrenia; Antipyretics Toxicity; Prolactin Excess
MeSH Terms: conditions — Schizophrenia; Hyperprolactinemia | interventions — Antipsychotic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: Antipsychotic — any antipsychotic medicine that would have the effect on prolactin level, such as amisulpride, risperidone, olanzapine and so on.

SUMMARY:
Objective:

Hyperprolactinemia(HPRL) which can result in a series of prolactin-related symptoms is a frequent adverse effect of antipsychotics. The investigators are interested to explicate the characteristics of serum prolactin level change after taking different antipsychotics and related factors.

Method:

1. Review of electronic medical records of schizophrenia patients who were brought to Shanghai Mental Health Center since January 1, 2007.
2. The investigators collect their information, and then

   1. set serum prolactin level after first 1-month antipsychotic treatment as primary outcome. Secondary outcomes are prolactin levels tested at other time points.
   2. Variables will range from antipsychotic kinds, dosage, treatment duration and blood concentration to demographic information, to disease history, to clinical treatment on hyperprolactinemia, to laboratory test results, such as blood routine examination, biochemistry, sex hormone levels and so on.
   3. After data cleaning and management, we will apply logistic regression, cox regression, Receiver Operating Characteristic curve (ROC) and machine learning to

      * analyze factors of prolactin level;
      * establish a model of prolactin change with time;
      * propose optimal monitoring time of prolactin according to prolactin change with time;
      * analyze correlation among antipsychotics, prolactin and clinical characters, for the purpose to supply objective evidence for antipsychotic treatment.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as schizophrenia according to Diagnostic and Statistical Manual of Mental Disorders(DSM)-5;
* were taking or going to take antipsychotics;
* have the results of serum prolactin level.

Exclusion Criteria:

* other mental disorder;
* suffered endocrinic diseases of pituitary or thyroid gland;
* suffered other organic brain diseases;
* have the history of tobacco or alcohol abuse, or psychoactive drug substance abuse.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with schizophrenia who were taking or going to take antipsychotic medicine.
Sampling Method: Non-Probability Sample
Enrollment: 10363 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
prolactin level at first 1-month antipsychotic treatment | at first 1-month antipsychotic treatment
  Serum prolactin level may change significantly after one month antipsychotic treatment.

SECONDARY OUTCOMES:
prolactin level at other time points | after 2-month, 3-month and half a year treatment with antipsychotics
  Different patients have different tendencies of prolactin, so collecting prolactin level at different time after exposed to antipsychotics is necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Huafang Li, MD, PhD, Principal Investigator — Shanghai Mental Health Center
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang L, Zheng Y, Huang J, Yu W, Zhou L, He L, Li Y, Hu H, Li G, Shen Y, Zhang J, Li H. Patterns of Serum Prolactin Elevation Associated with Nine Second-Generation Antipsychotics in a Large Cohort of Patients with Schizophrenia. CNS Drugs. 2025 Dec;39(12):1317-1330. doi: 10.1007/s40263-025-01216-1. Epub 2025 Aug 19. PMID 40830714